CLINICAL TRIAL: NCT04927260
Title: French Long Term Registry With Longitudinal Follow up of PDGFRA D842V-GIST Patients : AVapritinib Real-life observatTORy
Brief Title: French Long Term Registry With Longitudinal Follow up of PDGFRA D842V-GIST Patients
Acronym: AVIATOR2020
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Leon Berard (Other)
Collaborators: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: AVIATOR2020
Record Dates: First submitted 2021-06-02; First posted 2021-06-15 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: GIST; GIST, Malignant; PDGFR-Alpha D842V
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- COHORTE PROSPECTIF
  Interventions: Drug: Patient treated by Avapritinib in real life
- COHORTE RETROSPECTIF
  Interventions: Drug: Patient treated by Avapritinib in real life

INTERVENTIONS:
Drug: Patient treated by Avapritinib in real life — The patients included are treated with Avapritinib as part of their care. There is no change in treatment associated with this study.
  Patients must regularly complete various questionnaires: FACT-G, FACT-COG, and a neuropsychiatrist or a trained physician will give them the MoCA.

SUMMARY:
GIST are rare mesenchymal tumors of the gastrointestinal tract characterized by somatic mutations in the gene encoding the KIT (85%) or the PDGFRα (8%) protein. Treatment of localized forms relies on adequate surgery without tumor spillage and sometimes systemic treatment with imatinib according to risk of relapse defined by localization, tumor size and mitotic count, as well as mutational status. More than 40% of cases may recur and metastasize. Advanced and relapsing forms are currently treated with oral tyrosine-kinase inhibitors (TKI) of KIT and PDGFR such as imatinib (standard treatment), sunitinib (2nd line) and regorafenib (3rd line). Nevertheless, imatinib has little or no activity in patients harboring the D842V mutation in the exon 18 of PDGFRα (20% of gastric GIST, 6% of all GIST patients). Consequently, other therapeutic alternatives are needed.

Results from the phase I single-arm NAVIGATOR study show that avapritinib has significant efficacy in GIST patients with PDGFRα D842V mutation (ORR = 86 %). In France, an authorization for temporary use (ATUc) starting on September 21st, 2020 has been granted by the National Agency for Safety of Medicines and Health Products (ANSM). It allows the early availability of avapritinib in France while waiting for Market Authorization Approval (AMM). This ATUc is now being followed by a post-ATU period.

The objective of this real-life registry is to perform a long-term longitudinal follow up of PDGFRA D842V-mutated GIST patients and to collect effectiveness and safety data. It will be implemented in parallel to the post-ATUc period until June 2023.

Moreover, this registry fulfills the HAS's ("Haute Autorité de Santé") request regarding the Establishment of an exhaustive registry of patients with GIST, harboring the D842V / PDGFRA mutation in France. This registry will specifically describe:

* patient characteristics, in particular patient age, of the disease characteristics, previous treatments;
* the clinical course;
* the occurrence of adverse events / effects;
* and the therapeutic strategy (endpoint of treatment or continuation).

Data from the electronic health record (EHR) will be collected. Moreover, as per the ANSM's requirements, quality of life and cognitive function will be investigated using FACT-G, FACT-Cog and MoCA questionnaires.

Undesirable effects will be collected as well. Follow-up is envisioned for a minimum of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* I1. Adult (≥18 years old), male or female
* I2. Patient with a histologically or cytologically-confirmed diagnosis of unresectable or metastatic GIST harboring the D842V mutation in the PDGFRα gene
* I3. . Diagnosis date later than Jan 1st 2010
* I4. Non opposition to the use of her/his data

Exclusion criteria :

* E1. Patient not meeting all the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with GIST harboring a PDGFRa D842V mutation diagnosed from 2010 and treated with Avapritnib or not can be included.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | up to 48 months
  survival of patients treated with Avapritinib in real life according to overall survival.

SECONDARY OUTCOMES:
Progression Free Survival | after 12, 24 and 36 months
  according to RECIST criteria
Incidence of long-term responders | up to 48 months
  (>24 months)
Duration of treatment | up to 48 months
  duration in months
Safety: Nature of AEs | up to 48 months
  AEs graded using Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Safety : Frequency of AEs | up to 48 months
  AEs graded using Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Safety : Severity of AEs | up to 48 months
  AEs graded using Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Cognitive impairment in real-life according to MoCA questionnaires | Day 1, Day 15, Month 2, Month 3, Month 6, Month 12, Month 18, Month 24, Month 36
  Montreal Cognitive Assessment (MoCA)
Cognitive impairment in real-life according to FACT-Cog | Day 1, Day 15, Month 2, Month 3, Month 6, Month 12, Month 18, Month 24, Month 36
  Functional Assessment of Cancer Therapy - Cognitive Function
Quality of life in real-life according to FACT-G questionnaire | Day 1, Day 15, Month 2, Month 3, Month 6, Month 12, Month 18, Month 24, Month 36
  Functional Assessment of Cancer Therapy - General

CONTACTS AND LOCATIONS:
Overall Officials: MEHDI BRAHMI, Principal Investigator — Centre Leon Berard
Locations (7):
- France (7):
  - CHRU Besançon, Besançon
  - Insitut Bergonié, Bordeaux
  - CHU Clermont Ferrand, Clermont-Ferrand
  - Centre Léon Bérard, Lyon
  - Institut de Cancérologie de l'Ouest (ICO), Nantes
  - CHU Robert Debré, Reims
  - Institut Gustave Roussy, Villejuif